CLINICAL TRIAL: NCT04922060
Title: Evaluation of Cerebral Venous Return With Internal Jugular Vein Blood Flow in Gynecological Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, EMİNE ASLANLAR, Assistant professor, Selcuk University
Other Study IDs: EASLANLAR
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Internal Jugular Vein (IJV) Blood Flow in Gynecological Laparoscopic Surgery
Keywords: Laparoscopic surgery; cerebral venous drainage; internal jugular vein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The steep Trendelenburg position (STP) provides an advantage in laparoscopic procedures as it optimizes the surgical image. In laparoscopic operations, the need for CO2 pneumoperitoneum (PP), together with this non-physiological position, raises concerns about the patient's physiological homeostasis. Although most patients seem to tolerate the combination of STP and PP, this method carries risks of ICP (intracranial pressure) and brain perfusion. The head-down position increases arterial pressure as well as CVP, thereby disrupting cerebral venous drainage and increasing hydrostatic pressures in the cerebral vascular system. This increases cerebrovascular resistance and decreases cerebral blood flow by increasing ICP and cerebral edema. Systemic CO2 absorption from pneumoperitoneum causes hypercarbia. Hypercarbia can increase cerebral blood flow through cerebral vasodilation.

Seventy-four percent to 95% of cerebral venous drainage in the supine position is provided by IJVs. Studies have shown that IJVs, which are responsible for most cerebral venous drainage, exhibit changes in diameter and blood flow due to TP. These studies were generally conducted on moderate TP and on healthy volunteers. In this study, we aim to evaluate the effects of a steep Trendelenburg position (25°) and pneumoperitoneum on IJV blood flow in patients undergoing operation under general anesthesia

ELIGIBILITY:
Inclusion Criteria:

ASA I-II physical status age between 18 and 65 years planned gynecological laparoscopic surgery. -

Exclusion Criteria:

history of head and neck surgery history of cerebrovascular disease ASA III-IV physical status

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-II physical status, age between 18 and 65 years, and planned gynecological laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-08 (Estimated); Primary Completion 2021-06-24 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in internal jugular vein blood flow in laparoscopic gynecological cases | 90 minute
  to evaluate the effects of the pneumoperitoneum (PP) and steep Trendelenburg position (STP) on cerebral venous return with internal jugular vein (IJV) blood flow in gynecological laparoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: emine ASLANLAR, Principal Investigator — selcuk univercity medical faculty

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583
- [Result] Yeoh TY, Venkatraghavan L, Fisher JA, Meineri M. Internal jugular vein blood flow in the upright position during external compression and increased central venous pressure: an ultrasound study in healthy volunteers. Can J Anaesth. 2017 Aug;64(8):854-859. doi: 10.1007/s12630-017-0903-3. Epub 2017 Jun 2. PMID 28577164
- [Result] Uluer MS, Sargin M, Basaran B. Comparison of the effect of the right lateral tilt position and Trendelenburg position on the right internal jugular vein in healthy volunteers: A prospective observational study. J Vasc Access. 2019 Nov;20(6):672-676. doi: 10.1177/1129729819838169. Epub 2019 Apr 12. PMID 30977416
- [Result] Lee JG, Park HB, Shin HY, Kim JD, Yu SB, Kim DS, Ryu SJ, Kim GH. Effect of Trendelenburg position on right and left internal jugular vein cross-sectional area. Korean J Anesthesiol. 2014 Nov;67(5):305-9. doi: 10.4097/kjae.2014.67.5.305. Epub 2014 Nov 26. PMID 25473458
- [Result] Terai C, Anada H, Matsushima S, Shimizu S, Okada Y. Effects of mild Trendelenburg on central hemodynamics and internal jugular vein velocity, cross-sectional area, and flow. Am J Emerg Med. 1995 May;13(3):255-8. doi: 10.1016/0735-6757(95)90194-9. PMID 7755812
- [Result] Marcus HE, Bonkat E, Dagtekin O, Schier R, Petzke F, Wippermann J, Bottiger BW, Teschendorf P. The impact of Trendelenburg position and positive end-expiratory pressure on the internal jugular cross-sectional area. Anesth Analg. 2010 Aug;111(2):432-6. doi: 10.1213/ANE.0b013e3181e2fe41. Epub 2010 May 19. PMID 20484538
- [Result] Ishida S, Miyati T, Ohno N, Hiratsuka S, Alperin N, Mase M, Gabata T. MRI-based assessment of acute effect of head-down tilt position on intracranial hemodynamics and hydrodynamics. J Magn Reson Imaging. 2018 Feb;47(2):565-571. doi: 10.1002/jmri.25781. Epub 2017 Jun 3. PMID 28577333